CLINICAL TRIAL: NCT02131740
Title: Relationship Between Eye Rubbing and Transient Changes in Corneal Parameters in Healthy Volunteers: A Randomised-Controlled Trial
Brief Title: Eye Rubbing and Transient Change in Corneal Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sussex Eye Hospital (Other Government)
Responsible Party: Principal Investigator, Mayank A. Nanavaty, Consultant Ophthalmic Surgeon, Sussex Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 140622
Record Dates: First submitted 2014-04-30; First posted 2014-05-06 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Ectasia
Keywords: corneal; eye rubbing
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eye rubbing intervention (Experimental): eye rubbing performed for 1 minute in horizontal direction, clockwise rest for 5 seconds eye rubbing for a further 1 minute
  Interventions: Other: Eye rubbing
- No eye rubbing (Active Comparator): no eye rubbing - comparator
  Interventions: Other: No eye rubbing

INTERVENTIONS:
Other: Eye rubbing — eye rubbing for 1 minute in horizontal direction clockwise, 5 second rest & eye rubbing for a further 1 minute.
  Arms: Eye rubbing intervention
Other: No eye rubbing — This eye will not be rubbed
  Arms: No eye rubbing

SUMMARY:
This study addresses the research question:

How does eye rubbing affect corneal (clear part of eye) parameters in healthy volunteers

The study objectives are:

1. To determine the corneal changes following eye rubbing
2. To assess tear film changes following eye rubbing
3. To investigate if there is an association between eye rubbing and axial length of the eye.

DETAILED DESCRIPTION:
Background

A human eye has a front clear window called cornea. This cornea should ideally be spherical but in some subjects, this cornea gets deformed to a cone shape. This cone shaped cornea is called keratoconus. This keratoconus will cause blurring of vision which may require the use of a rigid contact lens or surgical intervention to improve vision. One of the etiological factors for keratoconus is eye rubbing. Eye rubbing is very common in subjects with eczema and other chronic allergic conditions. It is believed that constant eye rubbing every few minutes over years may lead to permanent changes to corneal curvature leading to formation of keratoconus.

It is known from previous studies that eye rubbing causes transient changes in the shape of the clear window of the eye, these changes are returned to baseline at 5 minutes following 1 minute of eye rubbing.

Although clinicians routinely advise such subject to refrain from eye rubbing and prescribe them long term anti allergic medication, there is paucity of scientific evidence on this.

With the knowledge of rubbing induced changes to the clear part of the eye in relation to the axial length we will have a further understanding of those subjects who are more susceptible to moulding and mechanical injury of the clear part of the eye. If we can identify a relationship between eye rubbing and eye length then those subjects with a chronic stimulus to eye-rubbing, such as allergy etc, efforts can be made to protect the eye from rubbing induced changes to prevent disease progression (Keratoconus).

The aim of this study is to assess transient changes (if any) in corneal and surface tear film parameters in healthy volunteers after rubbing of the right eye for 2 minutes. The volunteers will undergo a tear film assessment and a corneal scan before and after eye rubbing on both eyes. In addition to these, the volunteers will also undergo a simple scan (IOLMaster scan) to assess the overall dimension of their eyeballs before eye rubbing. The data from both eyes will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above healthy

Exclusion Criteria:

* aged less than 18 years
* subjects with: terminal illness, poor English language skills or a confused state history of previous ocular problems or surgeries history of contact lens wear not will to undergo simple & quick scans and eye examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
changes in corneal parameters following eye rubbing | pre and post eye rubbing for 2 minutes
  To study the change in anterior and posterior corneal parameters

SECONDARY OUTCOMES:
Relationship between eyeball dimensions following eye rubbing | pre and post eye rubbing for 2 minutes
  To study the relationship between the dimensions of the eye and the changes in corneal parameters following eye rubbing

CONTACTS AND LOCATIONS:
Overall Officials: Mayank Nanavaty, Consultant, Principal Investigator — Sussex Eye Hospital
Locations (1):
- Sussex Eye Hospital, Brighton, East Sussex, United Kingdom

REFERENCES:
- [Derived] Chervenkoff JV, Hawkes E, Ortiz G, Horney D, Nanavaty MA. A randomized, fellow eye, comparison of keratometry, aberrometry, tear film, axial length and the anterior chamber depth after eye rubbing in non-keratoconic eyes. Eye Vis (Lond). 2017 Aug 14;4:19. doi: 10.1186/s40662-017-0084-8. eCollection 2017. PMID 28815191